CLINICAL TRIAL: NCT00147485
Title: A Phase 1 Safety, Pharmacokinetic And Pharmacodynamic Study Of AG-024322, An Inhibitor Of Cyclin-Dependent Kinase 1, 2 And 4, Administered Intravenously Daily For 5 Days Every 3 Weeks To Patients With Advanced Cancer
Brief Title: A Phase 1 Study Of An Intravenously Administered Cyclin-Dependent Kinase Inhibitor In Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A7091001
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Neoplasms; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Neoplasms; Lymphoma, Non-Hodgkin | interventions — N-((5-(3-(4,6-difluoro-1H-benzimidazol-2-yl)-1H-indazol-5-yl)-4-methylpyridin-3-yl)methyl)ethanamine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AG-024322

INTERVENTIONS:
Drug: AG-024322

SUMMARY:
AG-024322 may work in cancer by stopping cancer cells from multiplying. AG-024322 is and intravenous drug from a new class of drugs call cyclin-dependent kinase (CDK inhibitors). This research study is the first time that AG-024322 will be given to people.

DETAILED DESCRIPTION:
The study was prematurely discontinued due to the inability of the compound to adequately differentiate from other treatment options in the clinical endpoint and necessary product profile on April 13, 2007. Safety profile was not the reason that led to the discontinuation of the program.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors or follicular of diffuse large cell non-Hodgkin's lymphoma, histologically or cytologically proven at diagnosis which is refractory to or intolerant of established therapy know to provide clinical benefit for their condition
* Adequate blood cell counts, kidney function and liver function and and ECOG score of 0 or 1.

Exclusion Criteria:

* Prior high-dose chemotherapy requiring hemapoietic stem cell rescue
* Previous radiation therapy to >25% of the bone marrow
* Active or unstable cardiac disease or history of heart attack within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To test the safety of AG-024322 when taken by people who have cancer
To find the AG-024322 dose that should be used in future clinical trials that will study effectiveness
To assess how the human body handles blood concentrations of AG-024322

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7091001&StudyName=A%20Phase%201%20Study%20Of%20An%20Intravenously%20Administered%20Cyclin-Dependent%20Kinase%20Inhibitor%20In%20Patients%20With%20Advanced%20Cancer